CLINICAL TRIAL: NCT01379443
Title: The Comparative Effect and Expense of More and Less Integration of Services That Provide Treatment and Rehabilitation for Children With Multiple Disabilities: A Randomized Controlled Trial
Brief Title: Rehabilitation of Children With Multiple Disabilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Treatment Network (Network)
Collaborators: McMaster University (Other)
Responsible Party: Sandy Thurston, Children's Treatment Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2008H00766
Record Dates: First submitted 2011-06-14; First posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Cerebral Palsy; Autism; Down's Syndrome; Brain Injury
Keywords: Children; Rehabilitation; Family Functioning; Mental Health; Costs; Integration
MeSH Terms: conditions — Cerebral Palsy; Autistic Disorder; Down Syndrome; Brain Injuries; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parental reports of their children (Active Comparator): Parental report of family-centered processes of care (MPOC) Parent mental health Parent perceived social support
  Interventions: Other: CTN model of care for children and their families
- Integration of service provider teams (No Intervention): Network co-alition teams were measured using the Integration of Human Services Measure, the Partnership Synergy Measure and a Network Capacity Measure were employed at the CEO level.

INTERVENTIONS:
Other: CTN model of care for children and their families — Parental reports on the quality of life of their children and service needs
  Arms: Parental reports of their children

SUMMARY:
The objective of the study is to compare the usual care and treatment of children and youth (0-19 years) with multiple developmental delays and disabilities and their families in Simcoe York with a co-ordinated, navigated approach to care using the Children's Treatment Network (CTN) services.

DETAILED DESCRIPTION:
The Children's Treatment Network (CTN)links existing children's services rather than creating a new Centre. The purpose of the evaluation is to compare the effectiveness and efficiency of this service with the usual care that people receive. 500 Children will be randomized to receive either usual care (250) or the co-ordinated, navigated care from CTN (250). The primary question to be addressed is whether the more integrated CTN model of service improves family-centered services, parent mental health, parenting, family function and the quality of the child's life and the families resource needs as well as reduce expenditures for the families' use of all other health and social services compared to the outcomes of usual care alone. What children and families with what characteristics and circumstances most benefit from which approach to the treatment of childhood disability in Simcoe-York? At what cost?

Agencies providing services to children will be evaluated as to how effective their integration of teams are functioning, their partnership with each other and capacity building in the community.

ELIGIBILITY:
Inclusion Criteria:

* Children and youth up to 19 years of age
* living in Simcoe-York.
* English speaking
* multi-need family
* children on agency service wait lists
* children under the care of Children's Aid Societies
* Families with more than 1 disabled child

Exclusion Criteria:

-youth over 19 years.

Ages: 1 Minute to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 445 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Parental reports in the Quality of Life of Children and Youth | 12 and 24 month
  Parent report of family centred processes of care (MPOC) Parent mental health Parent perceived social support

SECONDARY OUTCOMES:
Integration of teams amongst service providers. Integration was measured at two levels using the Integration of Human Services Measure. | 12 months and 24 months
  The measure evaluates observed and expected depth of integration among service providers.
  CEO or senior manager participation in the Network was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Thurston, Principal Investigator — Children's Treatment Network
Locations (1):
- McMaster University, Hamilton, Ontario, Canada